CLINICAL TRIAL: NCT00452907
Title: Assessment of the Public Health Benefit of Artemisinine Based Combination Therapies for Uncomplicated Malaria Treatment in Mali
Brief Title: ACT MALI: Treatment of Malaria Based on Combination Therapies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARTEN_L_00848
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Artesunate; sulfadoxine-pyrimethamine-artesunate; Lumefantrine

ARMS (3):
- 1 (Experimental): Arsucam® (AS 50mg/Aq153mg),oad, per os, 3 days of treatment
  Interventions: Drug: Artesunate
- 2 (Active Comparator): Arsumax (AS 50mg) + Sulfadoxine-Pyrimethamine (SP=SDX 500mg/PYR 25mg), oad, per os
  Interventions: Drug: Artesunate + Sulfadoxine-Pyrimethamine
- 3 (Active Comparator): Coartem (arthemether 20mg+ lumefantrine 120 mg), bid, per os. Duration of treatment: 3 days
  Interventions: Drug: arthemether + lumefantrine

INTERVENTIONS:
Drug: Artesunate — oad, per os, 3 days of treatment
  Arms: 1
Drug: Artesunate + Sulfadoxine-Pyrimethamine — oad, per os
  Arms: 2
Drug: arthemether + lumefantrine — bid, per os. Duration of treatment: 3 days
  Arms: 3

SUMMARY:
Test the hypothesis that repeated administration of Artesunate/Amiodaquine, Artesunate/Sulfadoxine-Pyrimethamine and Arthemeter-Lufemantrine for the treatment of consecutive episodes of uncomplicated malaria reduces the incidence of uncomplicated falciparum malaria and malaria attributable anemia

ELIGIBILITY:
Inclusion Criteria:

* Body weight > 5kg
* Residence in the investigator site area for the duration of the trial
* Axillary temperature ≥ 37,5°C at Day 0
* Confirmed Plasmodium falciparum infection,with parasitemia range from 2000 to 200000 asexual parasites /µl of blood

Exclusion Criteria:

* Danger signs or signs of severe malaria
* Other severe illnesses
* Allergy to one of the drugs
* Pregnant women

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 780 (Actual)
Dates: Start 2005-07; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Clinical and parasitological cure rate | at day 28
Clinical and biological tolerability | During the study period

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Lameyre, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bougoula, Mali